CLINICAL TRIAL: NCT06779955
Title: The Research Was Planned As a Randomized Controlled Experimental Study to Evaluate the Effects of Foot Massage on Back Pain and Vital Signs in Patients Undergoing Coronary Angiography.
Brief Title: Effect of Foot Massage After Coronary Angıography on Back Paın and Vıtal Sıgns
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ayşenur kahveci (Other)
Responsible Party: Sponsor-Investigator, ayşenur kahveci, PhD student and nurse, Cukurova University
Organization: Cukurova University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 0000-0003-2304-2994
Record Dates: First submitted 2024-12-18; First posted 2025-01-17 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Coronary Angiography (CAG)
Keywords: CAD; NURSİNG; ayak masajı

STUDY DESIGN:
Intervention Model Description: Simple randomization was used in the study.By computer randomization ,patients were divided into intervention and control groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- foot massage (Experimental): Pain and vital signs will be assessed for patients in the intervention group half an hour after they have stabilized after angiography. Foot massage will be applied at 1 hour after angiography. 8 minutes of foot massage will be applied to each foot (16 minutes in total for both feet). Vital signs and VAS will be assessed again immediately after the application, at 4 hours and at 8 hours.
  Interventions: Behavioral: foot massage application
- control group (No Intervention): No application will be made to the patients in the control group, and only the routine post-angiography care services of the service will be provided. Pain and vital signs assessment will be repeated half an hour, 1 hour, 4 hours and 8 hours after the patients leave the angiography.

INTERVENTIONS:
Behavioral: foot massage application — The characteristics of Massage Manipulations are an important feature in planning. Since the purpose of the massage is to rest, calm and relax, Effleurage (Stroke), Petrisage (Kneading) and Friction (Circular Rubbing) techniques that support circulation and have a loosening effect on the tissues have been chosen.A massage will be given to both feet for a total of 16 minutes, 8 minutes for each foot.The person receiving the massage will be lying down comfortably in a supine position, supported by pillows under the head and lower legs.Foot massage will be applied once to patients in the supine position at the first hour after their admission to the coronary intensive care unit following transfemoral angiography.
  Arms: foot massage

SUMMARY:
The aim of the study was to evaluate the effect of foot massage on patients' back pain and vital signs after coronary angiography. It is important for the transfer of nonpharmacological methods to clinical applications

DETAILED DESCRIPTION:
Cardiovascular diseases are the leading cause of death worldwide. According to the World Health Organization (WHO) data, approximately 393 million people lost their lives due to cardiovascular diseases in 2019. Similarly, when we look at the causes of death in our country, cardiovascular diseases are the leading cause.

Coronary artery disease (CAD), which is among the cardiovascular diseases, is the most important cause of mortality and morbidity. It is also one of the serious diseases that cause significant moral and financial burden on society . Sedentary lifestyle, change in eating habits, smoking, increased life expectancy with advancing technology, diabetes, hypertension and hyperlipidemia increase the prevalence of cardiovascular diseases. The increasing prevalence of risk factors among healthy individuals suggests that the material and moral burden caused by CAD will increase in the near future.

Early diagnosis and treatment are of vital importance in terms of prognosis in coronary artery diseases . Coronary angiography (CAG) is the gold standard in the diagnosis of CAD. Coronary angiography (CAG) and percutaneous transluminal coronary angioplasty (PTCA) are the most commonly used invasive procedures in the diagnosis and treatment of CAD. Complications frequently encountered after the CAG procedure are thromboembolism, bleeding, and hematoma. In order to prevent local vascular complications that may occur at the entry site after the TFA procedure, patients should lie flat in the supine position for approximately 4-8 hours after the procedure, depending on the protocols of each hospital. Although the flat supine position is considered safe, it causes various problems in patients. Studies have shown that lying flat on the back for a long time causes complaints such as orthostatic hypotension, aspiration risk, decreased oxygen saturation, urinary retention, increased cardiac load, and back pain. After coronary angiography, patients mostly complain of back pain, and the incidence of back pain has been reported to be between 11.4% and 26.5% .

Back pain can increase sympathetic stimulation, which can increase heart rate, blood pressure, cardiac load, and myocardial oxygen consumption. These problems contribute to worsening myocardial ischemia. Therefore, management of back pain after CAG is of great importance, especially in patients with serious cardiac problems. Pharmacological and non-pharmacological methods are used in pain management. Although painkillers are the most common pain relief method, they can cause side effects such as inadequate pain relief, respiratory depression, somnolence, nausea, vomiting, and paralytic ileus. Therefore, healthcare professionals frequently apply safer integrated health practices that can reduce pain without causing serious side effects. Integrative health practices such as distraction, music, acupressure, aromatherapy, acupuncture, transcutaneous electrical nerve stimulation (TENS), hot and cold applications and massage are used to reduce pain. Massage reduces pain by reducing cortisol and norepinephrine levels, increasing serotonin levels, stimulating endorphin release, facilitating blood flow, and increasing oxygenation in soft tissues. Another mechanism of action of massage is explained by the gate control theory, which argues that massage stimulates large nerve fibers and thus prevents pain signals from being transmitted to the central nervous system . There are many massage methods, such as whole-body massage, back massage, hand massage, and foot massage. Foot massage is among the most common types of massage. In foot massage, a certain amount of pressure is applied to certain points on the sole, which can affect the parts of the body associated with these points . Foot massage facilitates blood and lymph circulation in the body, thus accelerating the removal of waste products from the body, softening and stabilizing the movements of muscles, joints, and tendons, increasing muscle strength, and providing relaxation. Foot massage is a simple, inexpensive, and noninvasive procedure that can be used anywhere without the need for any special equipment and without compromising patient privacy. Kardan et al. In a study conducted by Kotrucihin et al., it was found that foot massage applied after coronary angiography reduced back pain.

Studies have reported that foot massage has positive effects on sleep quality, blood pressure and anxiety in patients with coronary disease, and that it reduces pain intensity and analgesic use when applied after surgery.

Pain diagnosis and control require teamwork. Within this team, nurses have an indispensable role as the healthcare personnel who spend the longest time with the patient. Relieving the patient's pain and increasing their comfort is an important part of nursing care. Nurses, who perform many applications while performing this task, also use massage, which is the most reliable pain control method.

The aim of this study was to evaluate the effect of foot massage on back pain and vital signs after CAG.

ELIGIBILITY:
Inclusion Criteria:

* Literate
* Over 18 years of age,
* Transfemoral CAG,
* No vision or hearing problems,
* Dorsal pedal and posterior tibial pulses are normal,
* No back pain in the last week before CAG,

Exclusion Criteria:

* No physiological or hemodynamic instability during and after CAG,
* Sensory disorders that impair the perception of back pain (paraplegia)
* Active bleeding at the site of cardiac dysrhythmia or catheter insertion,
* Known hemorrhagic disorders,
* History of spinal surgery or herniated disc in the lower back,
* Inflammation or infection in the leg or sole,
* Serious health problems in the feet,
* Not using opioid agents, tranquilizers or anesthetics before, during and 4 hours after CAG

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-01-15 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-10-15 (Estimated)

PRIMARY OUTCOMES:
Effect of foot massage after coronary angiography on back pain | The scale will be re-applied to patients half an hour, at the 1st hour, at the 4th hour and at the 8th hour after angiography.
  Visual Analog Scale, The scale was developed by Freyd M. in 2001. VAS, which is a simple, effective, repeatable and minimally instrumented measurement tool, is a one-dimensional scale frequently used in the measurement of subjective parameters. The scale consists of a 10 cm long line drawn vertically or horizontally. At both ends of this line are the two extreme descriptive words of the subjective category (0 = "no pain at all", 10 = worst/unbearable pain"). The patient is asked to mark the appropriate place on this line where the pain intensity will intersect. The distance from the lowest VAS level to the patient's mark is measured with a ruler and the numerical value of the patient's pain intensity is obtained in centimeters(cm) or millimeters (mm).
Effect of foot massage after coronary angiography on vital signs | The scale will be re-applied to patients half an hour, at the 1st hour, at the 4th hour and at the 8th hour after angiography.
  Vital Signs Evaluation Form:Pulse(bpm), systolic blood pressure (mmHg), diastolic blood pressure (mmHg) and respiratory rate measurements(breaths/minute) of the patients before and after the procedure will be recorded on the form prepared by the researcher.

CONTACTS AND LOCATIONS:
Locations (1):
- Çukurova Üniversitesi, Adana, Adana, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Pre- and post- implementation results of intervention and control group scales (statistical analysis). Participants' descriptive characteristics and participant consent form.
Supporting Information: ICF
Time Frame: Once published, the data is available indefinitely.
Access Criteria: Data can be shared publicly.
URL: https://tez.yok.gov.tr/UlusalTezMerkezi/